CLINICAL TRIAL: NCT04957056
Title: Finite Element Study of Biomechanical Changes After Unilateral Hemilamina and Facet Joint Resection of Cervical Spine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: M2018028
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Intraspinal Tumor
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study object: A young patient hospitalized in the Department of Neurosurgery of the Third Hospital of Beijing University of Medicine underwent CT examination of cervical vertebrae. The patient had no cervical bony deformity, no cervical degeneration, and no history of trauma
  Interventions: Procedure: Hospitalization

INTERVENTIONS:
Procedure: Hospitalization — Hospitalization

SUMMARY:
Finite element method was used to simulate unilateral hemilaminectomy of cervical spine and facet joint resection of different degrees, and the range of motion and the stress changes of ligament, intervertebral disc and endplate were calculated immediately after operation

DETAILED DESCRIPTION:
The finite element method was used to simulate unilateral hemilaminectomy of cervical spine and different degrees of facet joint resection, and the range of motion and the stress changes of ligaments, intervertebral discs and endplates were calculated immediately after the operation.

Finite element method was used to simulate unilateral hemilaminectomy of cervical spine and facet joint resection of different degrees, and the range of motion and the stress changes of ligament, intervertebral disc and endplate were calculated immediately after operation.

Study Design:

This study is a retrospective and general observational study.In this study, a young patient who was hospitalized in the Neurosurgery Department of the Third Hospital of Beijing University of Medicine and had undergone CT examination of cervical vertebra was selected. The patient had no cervical bony deformity, no cervical degeneration, and no history of trauma.

CT imaging data were collected, and a three-dimensional finite element model of C2-T1 segment of human cervical spine was established by finite element software. On the basis of this model, two and three levels of unilateral hemilamina and different degrees of facet joint resection were simulated.The lower end of the T1 vertebral body was fixed as the boundary condition, and three loading modes were adopted, namely, 2.0nm pure torque was applied to the upper surface of the C2 vertebral body along the sagittal plane, coronal plane and axial plane, respectively.The range of motion between vertebral segments was calculated and compared in different lamina surgical models. The tension of ligaments, the pressure of endplates and the pressure of intervertebral discs were obtained by finite element post-processing

ELIGIBILITY:
Inclusion Criteria:

A young patient hospitalized in the Department of Neurosurgery of the Third Hospital of Beijing University of Medicine underwent CT examination of cervical vertebrae.

Exclusion Criteria:

Cervical bony deformity Cervical degeneration History of trauma

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A young patient hospitalized in the Department of Neurosurgery of the Third Hospital of Beijing University of Medicine underwent CT examination of cervical vertebrae. The patient had no cervical bony deformity, no cervical degeneration, and no history of trauma
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Verification of the model | Through study completion, an average of 1 year
  In this study, the pure torque of 2.0Nm was applied to the upper surface of C2 vertebral body along the 1, 2 and 3 coordinates according to the right hand helical rule to generate the corresponding pure torque in the sagittal plane, coronal plane and axial plane, and to simulate the cervical spine flexion and extension, lateral bending and left-right rotation in real life

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Yu Wang, Study Chair — Peking University Third Hospital; Qi-Guo Rong, Study Director — Peking University
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No